CLINICAL TRIAL: NCT04549090
Title: Ultrasound Guided Posterior Quadratus Lumborum Block for Improved Postoperative Analgesia in Minimally Invasive Gynecologic Surgery
Brief Title: Ultrasound Guided Posterior Quadratus Lumborum Block for Postoperative Analgesia in Gynecologic Surgery
Status: Completed | Type: Observational
Sponsor: Pedram Bral (Other)
Responsible Party: Sponsor-Investigator, Pedram Bral, Principal Investigator, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2020-02-01
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Post-operative Pain; Gynecologic Surgery; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- No QL block group: These patients will not be receiving QL block based on their shared decision with their surgeon and anesthesiologist. Patients' pain scores and amount of pain killers will be followed up for 24 hours postoperatively
- QL block group: These patients will be receiving QL block based on their shared decision with their surgeon and anesthesiologist. Patients' pain scores and amount of pain killers will be followed up for 24 hours postoperatively
  Interventions: Drug: QL (quadratus lumborum) block administration

INTERVENTIONS:
Drug: QL (quadratus lumborum) block administration — Fo the QL block group, they will be receiving bilateral QL block. A total of 40ml of 0.25% bupivacaine (Marcaine) and 10ml of liposomal bupivacaine (Exparel) will be administered
  Groups: QL block group

SUMMARY:
The challenge to achieve adequate analgesia has led to the development of directed, multi-modal protocols specific to management of post-laparoscopy pain in effort to decrease the amount of additional administration of narcotic medication. While several non-opioid regiments have been found to be effective, opioid medications still play a significant role in early postoperative analgesia. Given the adverse side effects of narcotic medications, regional blocks utilizing local anesthetic agents and has been shown to improve overall pain control in this time period.

Truncal abdominal nerve blocks are useful for pain control in abdominal and pelvic surgeries. More recently, the utilization of the quadratus lumborum (QL) block has effectively alleviated somatic and visceral pain in the upper and lower abdomen. The QL block provides analgesia spanning from the T4 to L1 dermatomal levels in the thoracolumbar plane to provide a broad sensory level analgesic effect. The approach involves injecting local anesthetic under ultrasound guidance into the plane posterior to the quadratus lumborum muscle and middle layer of thoracolumbar fascia.

Given the utility of the QL block in controlling somatic pain, this study aims to determine whether the QL block is an effective analgesic adjunct in the control of postoperative pain period, specifically with regards to patients undergoing laparoscopic gynecologic surgery.

DETAILED DESCRIPTION:
Prospective Cohort observational study. All patients that meet criteria for participation in this study will be screened: patients scheduled to undergo a laparoscopic hysterectomy for benign conditions by attending physicians in the division of Minimally Invasive Gynecologic Surgery. Based on surgeon's preference, and patient's consent, the patient is offered a QL block or not. Our aim is to follow the patient's pain scores post op and amount of oral pain medication used whether they received QL block or not. If the patient received the QL block then they will be considered part of the study arm. If the patient did not receive the QL block then they will be considered part of the control arm.

The QL block is best thought of as a volume or compartment block in that volumetric spread of LA along the fascial plane is associated with efficacy in blocking the thoracolumbar nerves between T7-L1. It can be reasonably assumed that this compartment is the same across patients and is not affected by the amount of subcutaneous or central fat present in the obese patient.

If a block is to be performed, the QL block will be performed using a 21G x 100mm Stimuplex needle under ultrasound guidance using a curvilinear probe. Subjects will be positioned in the semi-lateral position to facilitate access into the plane posterior to the quadratus lumborum muscle and middle layer of thoracolumbar fascia. The QL block will be administered via an in-plane approach and local anesthetic will be injected between the quadratus lumborum muscle and the middle layer of the thoracolumbar. The QL block will be in the operating room after induction prior to starting the scheduled surgical procedure. If the block is performed, it will include 20ml of 0.25% bupivacaine and 5ml of liposomal bupivacaine (Exparel) per side. The block will be done bilaterally therefore a total of 40ml of 0.25% bupivacaine and 10ml of liposomal bupivacaine (Exparel) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for recruitment if between the ages of 18 to 65 scheduled to undergo laparoscopic or robotic total or supracervical hysterectomy for benign indications. Only surgery for benign pathology will be considered to enrollment. No Malignancy cases will be included.

Exclusion Criteria:

* 1. History of adverse reaction or allergy to Bupivacaine or liposomal bupivacaine

  2. Medical contraindication to placement of QL block.

  3. Suspicion of possible reproductive cancer with contraindication of morcellation of uterine tissue.

  4. Significant medical condition or laboratory result that in the opinion of the Investigator indicate an increased vulnerability to study subject which exposes the subject to an unreasonable risk as a result of participating.

  5. Any clinically significant condition uncovered during the surgery, such as excessive bleeding or decompensation, that might render the subject medically unstable to continue the study or complicate the subject's intraoperative or postoperative course.

  6. Pregnant patients

  7. Less than 40Kg weight.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 to 65 scheduled to undergo laparoscopic or robotic total or supracervical hysterectomy for benign indications
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Difference in pain score | 3 hours postoperative
  Our primary outcome is difference in pain scores at 3 hours between the two groups. The pain score will be assessed using Numeric Rating Scale (NRS) from 0-10 with 0 as no pain and 10 as worst possible pain

SECONDARY OUTCOMES:
Difference in pain score | 1 hour postoperative
  Our secondary outcome is difference in pain scores at 1 hour between the two groups. The pain score will be assessed using Numeric Rating Scale (NRS) from 0-10 with 0 as no pain and 10 as worst possible pain
Difference in pain score | 24 hours postoperative
  Our secondary outcome is difference in pain scores at 24 hour between the two groups. The pain score will be assessed using Numeric Rating Scale (NRS) from 0-10 with 0 as no pain and 10 as worst possible pain
Difference in amount of pain killers used | pain killers used during the 24 hours postoperatively. The patient will be provided an empty sheet to record everytime a pain killer is used including the type and dose of pain killer . The pain killers are prescribed at the surgeon's discretion
  Our secondary outcome is difference in the amount of pain killers used during the 24 hour period post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Bral, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT04549090/Prot_SAP_000.pdf